CLINICAL TRIAL: NCT03471286
Title: A Phase 1b Window of Opportunity Study to Investigate Mechanisms of Actions of Novel Therapeutic Agents in Patients With Resectable Solid Tumor Malignancies
Brief Title: A Window of Opportunity Study to Investigate Mechanisms of Actions of Novel Therapeutic Agents in Patients With Resectable Solid Tumor Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Deprioritization of drug in this patient population
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J17168; IRB00156271 (Other: JHM IRB); I-24360-17-13 (Other: Incyte Corporation)
Record Dates: First submitted 2018-03-02; First posted 2018-03-20 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Solid Tumor
MeSH Terms: interventions — epacadostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sub-Protocol A (Experimental): Epacadostat
  Interventions: Drug: Epacadostat

INTERVENTIONS:
Drug: Epacadostat — Drug is taken orally two times per day for 14 days, prior to surgical resection of tumor.

SUMMARY:
This is a single-institution, single arm, open label, window of opportunity clinical trial that will act as a Master Protocol with a primary objective to assess pharmacodynamic effects of the novel study drugs in subjects with resectable solid tumor malignancies.

Each Sub-protocol conducted under the Master Protocol will evaluate different novel therapeutic agent(s).

Estimated enrollment is 15 subjects per Sub-Protocol.

DETAILED DESCRIPTION:
Patients will have a short-course (4-weeks) administration of a given compound in the timeframe between the diagnostic biopsy and the surgical resection. A pre-treatment tumor biopsy will be obtained, and blood samples will be collected before, during, and at the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Must have biopsy-proven solid tumor that is eligible for elective surgical resection, disease does not require immediate therapy, and there is NO approved/ standard therapy available that is shown to prolong overall survival.
2. ECOG performance status of 0 or 1.
3. Must have a tumor lesion that is amenable to biopsy, and willing to undergo biopsy.
4. Willing to provide tissue and blood samples for research.

Exclusion Criteria:

1. The following solid tumors are NOT eligible: Primary brain tumor, Ocular melanoma, Head and neck cancer, Breast cancer, Prostate cancer, Testicular cancer, and Stage III rectal cancer.
2. Any active malignancy within 3 years prior, except: Adequately treated basal cell or squamous cell skin cancer, or early stage cancers (carcinoma in situ or stage 1) treated with curative intent.
3. Any uncontrolled intercurrent illness, including but not limited to: Symptomatic congestive heart failure, Unstable angina pectoris or coronary angioplasty or stenting within 6 months prior to enrollment, Cardiac arrhythmia, Psychiatric illness or social situations that would limit compliance with study requirements, or Ongoing or active infection.
4. Any known sensitivity to or history of allergic reaction to compounds of similar chemical or biological composition of study drug(s).
5. Unwilling or unable to follow the study schedule.

Other protocol defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-06-06 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamic effects as measured by changes in biomarkers in pre- and post-dose tumor and blood specimens | Approximately 1 year
  To establish baseline levels and measure pharmacodynamic biomarker changes in tumor and/or blood samples after treatment with the study drug.
  Sub- Protocol A will focus on changes in CD8+ T cells, CD4+Foxp3+ cells, NK cells, DCs and immune checkpoints.

SECONDARY OUTCOMES:
Safety and tolerability as measured by incidence of AEs (Adverse Events) | Approximately 1 year
  To assess the safety and tolerability of the study drug in the pre-surgical setting graded according to Common Terminology Criteria for Adverse Events (CTCAE), version 4.0.
Pathological Response Rate as measured by correlation of biomarkers in tumor and/or blood specimens | Approximately 1 year
  To evaluate pathological response rate of solid tumor malignancies in subjects receiving neo-adjuvant treatment with the study drug and to assess a possible correlation with biomarkers either in the tumor specimens either in the bloods samples and the pathological response.
Overall Survival | Approximately 2 years
  To determine the overall survival (OS) status of subject treated which the study drug at 6 months, 1 year and 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Nilofer Azad, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No